CLINICAL TRIAL: NCT04357145
Title: The Effect of Different Exercise Dosages on Exercise Adherence, Pain and Functionality in Patients With Knee Osteoarthritis
Brief Title: Exercise Dosages and Exercise Adherence With Patients With Knee Osteoarthritis
Acronym: Adherence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Eda Tonga, Doctor of Philosophy, Marmara University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 563254
Record Dates: First submitted 2020-04-20; First posted 2020-04-22 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Knee Osteoarthritis
Keywords: Knee Osteoarthritis; Exercise Adherence; Exercise Dosage; Home Exercises
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Exercise Group (Active Comparator): Exercise training is given to patients in the form of a home exercise program.
  Interventions: Other: Standard Dosage Home Exercise Training
- High Dosage Exercise Group (Experimental): The high dosage exercise training group will implement the recommended exercise program 3 times more than the standard exercise group.
  Interventions: Other: High Dosage Home Exercise Training

INTERVENTIONS:
Other: High Dosage Home Exercise Training — By giving more exercise to the experimental group, exercise adherence, pain and functionality will be compared with the standard exercise group.
  3 times more reputation than control
  Exercise Program to be Applied (0-3 Weeks):
  Isometric knee extensor and adductor exercise
  * Hamstring stretching exercise
  * Terminal knee extension exercise
  * Straight leg lifting exercise
  Exercise Program to be Applied (3-12 Weeks):
  * Stepping exercise
  * Sit up and stand up without support
  * Active knee flexion exercise
  * Moving forward exercise
  Arms: High Dosage Exercise Group
Other: Standard Dosage Home Exercise Training — 5-6 standard reputations for all exercises
  Exercise Program to be Applied (0-3 Weeks):
  Isometric knee extensor and adductor exercise
  * Hamstring stretching exercise
  * Terminal knee extension exercise
  * Straight leg lifting exercise
  Exercise Program to be Applied (3-12 Weeks):
  * Stepping exercise
  * Sit up and stand up without support
  * Active knee flexion exercise
  * Moving forward exercise
  Arms: Standard Exercise Group

SUMMARY:
Although the effects of different exercise dosages for patients with osteoarthritis are compared in the literature, it is seen that studies on which exercise dosage is better are insufficient.The planned study has 2 main objectives:

* To examine the effects of different exercise dosages on exercise dependence
* To investigate the effect of different exercise dosages on pain and functional results

DETAILED DESCRIPTION:
Knee osteoarthritis (KO) is the most common musculoskeletal problem worldwide, leading to pain and loss of locomotor function. The Framingham Osteoarthritis Study shows that 19% of adults have radiographic effects on the knee joint. Individuals with advanced symptomatic KO have difficulties in their daily life activities. Among all diseases, KO most affects activities such as walking, climbing stairs and housework. A wide range of physiotherapy treatment methods are available in KO treatment such as strengthening exercises, aquatic exercises, aerobic exercises, proprioception exercise, orthotics, taping methods and the use of electrophysiological agents. High-quality evidences suggests that land-based exercise therapy maintains its positive effect on pain, quality of life and functionality for 2-6 months after the treatment. The dosage of exercise therapy can be adjusted by the duration, frequency, or resistance of the exercise. However, evidence-based information on exercise dosage is limited in KO treatment. While KO is treated in physiotherapy clinics, it is also supported by home exercises during and after treatment. However, it is a clinical problem that patients show low adherence to home exercise. With this study, it is aimed to compare the exercise adherence of patients who are given home exercise with different exercise dosages and to show their functional results. Participants with KO aged between 40-85 years will be included in the study and randomly divided into two groups. The number of repetitions of the high dosage exercise group will be 2 times more than standard exercise group. Participants will be asked to apply home exercise programs 4 times a week. Exercise adherence, pain, kinesiophobia and functionality will be evaluated. Our study will be the first to demonstrate the effect of different home exercise dosages on exercise adherence. The information to be obtained with this study is thought to contribute to the preparation of a better home exercise program. With the information to be obtained through this study, it can contribute to the preparation of a better home exercise program.The planned study has 2 main objectives:

* To examine the effects of different exercise dosages on exercise dependence
* To investigate the effect of different exercise dosages on pain and functional results

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnosis of unilateral or bilateral knee osteoarthritis.
* Being between stage 1-3 according to Kellgren-Lawrence criteria.
* Having at least 3 months of pain duration and decreased functioning.
* Being a volunteer who can read and write

Exclusion Criteria:

* Physiotherapy or other conservative therapy during the previous 3 months or a history of major knee trauma.
* Having Inflammatory joint disease, hip symptoms more aggravating than the knee symptoms,
* Having comorbidities not allowing exercise such as cardiovascular, respiratory, systemic, or metabolic conditions limiting exercise tolerance.
* Participants with previously performed knee replacement surgery

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-10-30 (Estimated)

PRIMARY OUTCOMES:
Change from Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Points at 12 weeks | Baseline, Week 3, Week 6 and Week 12
  (WOMAC) is a widely used, proprietary set of standardized questionnaires used by health professionals to evaluate the condition of patients with osteoarthritis of the knee and hip, including pain, stiffness, and physical functioning of the joints.The WOMAC measures five items for pain (score range 0-20), two for stiffness (score range 0-8), and 17 for functional limitation (score range 0-68). Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
Change from Exercise Adherence (with Self Reported Exercise Diary) at 12 Weeks Percentages at 12 Weeks | Week 3, Week 6, Week 9, Week 12
  In the exercise diary, the participant will note the number of exercises done at home next to the image showing the exercise example day by day.The percentage adherence to the prescribed exercise regimen was calculated by dividing the number of exercises performed by the number of exercises prescribed and multiplying by 100.
Change from Knee Osteoarthritis Exercise Adherence Scale Points at 12 Weeks | Week 3, Week 6, Week 9, Week 12
  It consists of four yes / no questions.'Yes' answer is rated with 1 point, 'No' answer gets 0 point. Lesser scores indicate good exercise adherence.

SECONDARY OUTCOMES:
Change from Visual Analogue Scale(for Pain) Points at 12 Weeks | Baseline, Week 3, Week 6 and Week 12
  The pain Visual Analogue Scale(VAS) is a unidimensional measure of pain intensity, which has been widely used in diverse adult populations. VAS is a straight horizontal line of fixed length, usually 100 mm. The ends are defined as the extreme limits of the parameter to be measured pain orientated from the left (worst) to the right (best).
Change from Tampa Scale for Kinesiophobia Points at 12 Weeks | Baseline, Week 3, Week 6 and Week 12
  The term kinesiophobia refers to a fear of pain with movement - i.e., movements which a patient is hesitant to perform due to fear that the movement will elicit pain. Likert scoring with 4 points (1 = Strongly disagree, 4 = I totally agree) is used in the scale. Tampa Scale for Kinesiophobia consists of 17 questions. A score of 17 is the lowest possible score, and indicates no kinesiophobia or negligible. A score of 68 is the highest possible score and indicates extreme fear of pain with movement. A total score is calculated after inversion of the individual scores of items 4, 8, 12 and 16.
Change from Timed Up&Go Test Score at 12 Weeks | Baseline, Week 3, Week 6 and Week 12
  The timed up and walk test(TUG) is used to measure the time it takes for the patient to get up from the chair, walk a distance of 3m, turn and sit on the same chair. TUG is a simple test used to assess a person's mobility and requires both static and dynamic balance. One source suggests that scores of ten seconds or less indicate normal mobility, 11-20 seconds are within normal limits for frail elderly and disabled patients, and greater than 20 seconds means the person needs assistance outside and indicates further examination and intervention.
Change from Timed 10 Meter Walk Test Score at 12 Weeks | Baseline, Week 3, Week 6 and Week 12
  The 10 Metre Walk Test is a performance measure used to assess walking speed in metres per second over a short distance. It can be employed to determine functional mobility, gait, and vestibular function. The participant walks without assistance for 10 metres, with the time measured for the intermediate 6 metres to allow for acceleration and deceleration.

IPD SHARING:
Plan to Share IPD: No